CLINICAL TRIAL: NCT02631499
Title: Post-hepatectomy Adjuvant Transcatheter Arterial Chemoembolization for Hepatocellular Carcinoma Patients With Preoperative CTC Level ≥2: a Multicenter Randomized Controlled Trial in China
Brief Title: Efficacy Study of TACE to Treat Hepatocellular Carcinoma After Operation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Johnson & Johnson Medical, China (Industry)
Responsible Party: Principal Investigator, Jia Fan, President of Shanghai Zhongshan Hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC-HE-TACE
Record Dates: First submitted 2015-12-09; First posted 2015-12-16 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma, Hepatocellular; Neoplastic Cells, Circulating
Keywords: Circulating Tumor Cells; Hepatoectomy; TACE; prognosis; relapse; Chemoembolization, Therapeutic
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplastic Cells, Circulating; Recurrence | interventions — Chemoembolization, Therapeutic; Epirubicin; Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjuvant TACE (Experimental): TACE will be performed 4-6 weeks after hepatectomy in patients with preoperative CTC ≥2 Epirubicin, lipiodol and gelatin sponge articles are used in TACE.
  Interventions: Procedure: TACE; Drug: Epirubicin; Drug: lipiodol
- Control (No Intervention): no interventions were assigned after hepatectomy

INTERVENTIONS:
Procedure: TACE — TACE is performed 4-6 weeks after hepatectomy. Epirubicin and lipiodol are used in TACE.
  Other Names: Transcatheter Arterial Chemoembolization; Chemoembolization
  Arms: Adjuvant TACE
Drug: Epirubicin — Epirubicin is a chemotherapy drug used in TACE
  Other Names: EADM
  Arms: Adjuvant TACE
Drug: lipiodol — lipiodol is a kind of embolization material used in TACE
  Other Names: Ultra-fluid lipiodol
  Arms: Adjuvant TACE

SUMMARY:
This study is designed to prospectively evaluate whether post-hepatectomy adjuvant transcatheter arterial chemoembolization (TACE) is effective in reducing early recurrence in HCC patients with preoperative CTC ≥2.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most prevalent malignancies worldwide, and associated morbidity and mortality rates have escalated in recent years. Despite improvements in surveillance and clinical treatment strategies, the prognosis of HCC remains very poor due to high incidence of recurrence and metastasis. Recent clinical studies have provided evidence that circulating tumor cell (CTC) may directly participate in the metastasis cascade in various types of malignancies. The investigators previous data indicated that HCC patients with preoperative CTC levels ≥2 suffered significantly earlier recurrence (within 1 year) than patients with lower levels. However, the benefits of postoperative adjuvant therapies in preventing early recurrence in patients with preoperative CTC ≥2 remain to be elucidated. Transarterial chemoembolisation (TACE) is an effective palliative treatment for HCC. The investigators design a randomised controlled trial evaluating the efficacy of using TACE after hepatectomy to reduce early recurrence rates in HCC patients with preoperative CTC level ≥2.

ELIGIBILITY:
Inclusion Criteria:

* HCC patients received curative hepatectomy with negative resection margin
* Age from 18 to 75
* Child-Pugh class A
* ASA class I to II
* ECOG performance status Grade 0 or 1
* Preoperative CTC level ≥2 per 7.5 ml peripheral blood
* No residual tumor revealed by hepatic arterial angiography 4-6 weeks after hepatectomy

Exclusion Criteria:

* Patients diagnosed with other types of malignancies besides HCC
* Patients receiving concomitant local ablation or previous TACE
* Main portal vein tumor thrombus extraction during hepatectomy
* Hepatic arterial angiography before adjuvant TACE treatment reveals residual tumors.
* Presence of extra-hepatic or lymphatic metastasis
* Impaired liver function with either clinically detected ascites, hepatic encephalopathy, serum albumin < 25g/L or bilirubin > 50micromol/L
* Renal impairment with creatinine > 200micromol/L
* Severe concurrent medical illness persisting > 6 weeks after hepatectomy
* History of other cancer
* Hepatic artery anomaly making TACE not possible
* Allergy to 5-Fluorouracil, Epirubicin or lipiodol
* Pregnant woman
* Informed consent not available

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Early recurrence rates | 1 year after hepatectomy
  Early recurrence was defined as any type of recurrence diagnosed within 1 year after hepatectomy.

SECONDARY OUTCOMES:
Overall Survival | up to 3 years
  OS was defined as the interval from date of HCC resection to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD & PhD, Principal Investigator — Shanghai Zhongshan Hospital, Fudan University
Locations (6):
- China (6):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Eastern Hepatobiliary Surgery Hospital, Second Military Medical University, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Affliated with Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sun YF, Xu Y, Yang XR, Guo W, Zhang X, Qiu SJ, Shi RY, Hu B, Zhou J, Fan J. Circulating stem cell-like epithelial cell adhesion molecule-positive tumor cells indicate poor prognosis of hepatocellular carcinoma after curative resection. Hepatology. 2013 Apr;57(4):1458-68. doi: 10.1002/hep.26151. Epub 2013 Mar 4. PMID 23175471
- [Background] Zhong C, Guo RP, Li JQ, Shi M, Wei W, Chen MS, Zhang YQ. A randomized controlled trial of hepatectomy with adjuvant transcatheter arterial chemoembolization versus hepatectomy alone for Stage III A hepatocellular carcinoma. J Cancer Res Clin Oncol. 2009 Oct;135(10):1437-45. doi: 10.1007/s00432-009-0588-2. Epub 2009 May 1. PMID 19408012
- [Background] Ren ZG, Lin ZY, Xia JL, Ye SL, Ma ZC, Ye QH, Qin LX, Wu ZQ, Fan J, Tang ZY. Postoperative adjuvant arterial chemoembolization improves survival of hepatocellular carcinoma patients with risk factors for residual tumor: a retrospective control study. World J Gastroenterol. 2004 Oct 1;10(19):2791-4. doi: 10.3748/wjg.v10.i19.2791. PMID 15334671